CLINICAL TRIAL: NCT04431232
Title: Endoscopic Band Ligation for Weight Loss
Brief Title: Endo-Band: Endoscopic Band Ligation for Weight Loss
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: El Katib Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Abeid, Consultant Gastroenterologist/ Bariatric Endoscopist Cairo University, El Katib Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MohamedAbeid1
Record Dates: First submitted 2020-05-28; First posted 2020-06-16 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Obesity
Keywords: Obesity; BMI
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Band Ligation (Experimental): Band ligation of gastric body for weight loss
  Interventions: Device: Endoscopic Band Ligation

INTERVENTIONS:
Device: Endoscopic Band Ligation — Band ligation of the gastric body for weight loss

SUMMARY:
To the best of our knowledge, this is the first study to use endoscopic band ligation for weight loss. All ligatures will be performed in the gastric body starting at the distal body; 5 parallel rows, with the last one in the proximal body.The entire procedure can be completed in 30 min. Oxygen is used for endoscopic air insufflation.Endoscopy is performed using propofol for sedation.

DETAILED DESCRIPTION:
The idea of band ligation of the gastric body is to induce multiple gastric ulcers that forms a fibrotic scars which can lead to marginal narrowing of the lumen; same as that occurred in the esophagus following band ligation of esophageal varices or in the antrum following band ligation of GAVE.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 27

Exclusion Criteria:

* Any contraindication for endoscopy
* Any gastric bleeding lesions
* Uncontrolled use of anticoagulants or NSAID's

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-03-07 (Estimated); Study Completion 2026-03-07 (Estimated)

PRIMARY OUTCOMES:
Weight Loss | 3 months
  BMI Change

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abeid, MD, Principal Investigator — Endoscopy Unit Faculty of Medicine Cairo University
Locations (1):
- El Katib Hospital (Celopatra Group), Giza, Dokki, Egypt

REFERENCES:
- [Background] Keohane J, Berro W, Harewood GC, Murray FE, Patchett SE. Band ligation of gastric antral vascular ectasia is a safe and effective endoscopic treatment. Dig Endosc. 2013 Jul;25(4):392-6. doi: 10.1111/j.1443-1661.2012.01410.x. Epub 2012 Dec 17. PMID 23808945
- [Background] Jirapinyo P, Thompson CC. Endoscopic gastric body plication for the treatment of obesity: technical success and safety of a novel technique (with video). Gastrointest Endosc. 2020 Jun;91(6):1388-1394. doi: 10.1016/j.gie.2020.01.030. Epub 2020 Jan 28. PMID 32001332
- [Background] Abeid M, Miller KA, Kaddah T, Zaitoun N. Outcome of Primary Obesity Surgery Endolumenal Procedure as Obesity Treatment in Private Practice Setting: an Intervention Study. Obes Surg. 2019 Apr;29(4):1364-1366. doi: 10.1007/s11695-018-03698-z. No abstract available. PMID 30627991